CLINICAL TRIAL: NCT04472637
Title: Atorvastatin Effects On Arterial Stiffness In Hemodialysis Patients
Brief Title: Atorvastatin Effects On Arterial Stiffness In Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: arterial stiffness in HD
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Arterial Stiffness
Keywords: statin, hemodialysis
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: This research is a double-blinded , placebo-controlled, randomized clinical trial. Fifty patients with end-stage renal disease (ESRD) receiving hemodialysis treatment will be enrolled in the study.
  Patients will be randomly assigned using block randomization method into two study groups:
  Experimental group (25 patients): They will receive atorvastatin 10 mg, as one tablet /day for 24 weeks.
  Control group (25 patients): They will receive a placebo in the form of multivitamin tablets similar to the experimental drugs with the same regimen (one tablet /day for 24 weeks).
  Allocation concealment: will be ensured using sealed closed envelop randomization technique, every patient will be given an identification code.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: a double blinded study as participants, health care providers as well as the outcome assessor will be unaware about the type of treatment each patient receive.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): They will receive atorvastatin 10 mg, as one tablet /day for 24 weeks.
  Interventions: Drug: Atorvastatin
- placebo (Placebo Comparator): They will receive a placebo in the form of multivitamin tablets similar to the experimental drug with the same regimen, as one tablet /day for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 10 mg, as one tablet /day for 24 weeks.
  Other Names: Lipitor, Ator
  Arms: Atorvastatin
Drug: Placebo — a placebo in the form of multivitamin tablets similar to the experimental drugs with the same regimen (one tablet /day for 24 weeks)
  Arms: placebo

SUMMARY:
This research aims to assess effects of atorvastatin on arterial stiffness in hemodialysis patients

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the most common cause of morbidity and mortality among patients with end-stage renal disease (ESRD) on hemodialysis (HD).

CVD are present since the early stages of chronic kidney disease (CKD) and reach around 30 to 44% of those beginning hemodialysis. Macrovascular disease develops rapidly in uremic patients and is responsible for the high incidence of ischemic heart disease, left ventricular (LV) hypertrophy, congestive heart failure, sudden death, and stroke.

Compared with the general population, the incidence of cardiovascular (CV) events among patients with ESRD is significantly higher, but it does not seem to be fully explained by the increased incidence of conventional risk factors alone. It has been hypothesized that HD patients are exposed to unique renal and HD-related risk factors that predispose them to an increased rate of CV events. Research efforts have expanded understanding of the contribution made by vascular pathologies to this burden.

Clinicians now recognize that defects in the vascular wall are the bases of many CV events, and early detection and intervention in subclinical vascular disease are fundamental for preventing and controlling cardiovascular events. Changes in the vasculature include endothelial dysfunction (ED), smooth muscle cell hyperplasia/hypertrophy, vascular calcification, and arterial stiffness.

Arterial stiffness is one of the vascular pathologies in HD patients. Recent studies examining cardiovascular complications in dialysis patients focused on atherosclerosis, including arterial stiffness and wall thickness changes as a major contributing factors for CV events. It was shown that stiffening of arteries is associated with increased cardiovascular mortality and morbidity.

Arteriosclerosis refers to the reduced arterial compliance due to increased fibrosis, loss of elasticity, and vessel wall calcification affecting the media of large and middle-sized arteries. These arterial wall changes are influenced not only by nonspecific factors, such as age, genetics, hypertension, diabetes, lipid abnormalities, inflammation, and/or common atherosclerosis, but also by parameter(s) associated with the presence of uremia per se.

Arterial stiffening in patients with CKD and ESRD occurs at an accelerated rate compared with the normal ageing process and arteriosclerosis. As bone mineral metabolism worsens with advancement to ESRD, hyperphosphatemia, secondary hyperparathyroidism and inhibited vitamin D synthesis result in vascular calcification that causes hardening of the arteries. Other factors linked to the uremic environment, such as anaemia, endothelial dysfunction, neuro-hormonal activation and inflammation, play important roles.

Arterial stiffness can be assessed noninvasively with the use of pulse wave velocity (PWV) measurement. The aortic pulse wave velocity (APWV) reflects central arterial stiffness. APWV is a predictor of cardiovascular outcome in patients with hypertension, diabetes, end-stage renal disease, and elderly hospitalized subjects.

Statins or 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors are considered first-line treatment for elevated low-density lipoprotein cholesterol (LDL-C) levels, as large-scale, randomized clinical trials have demonstrated their clinical benefits in primary and secondary prevention of cardiovascular events. Background and clinical studies have also shown beneficial actions of statins for the vasculature that may extend above their lipid lowering properties, such as improvement of endothelial function, inhibition of vascular smooth muscle cell proliferation, and reduction of vascular inflammation. It has been also proposed that such pleiotropic effects of statins may translate into a beneficial impact on arterial stiffness. Atorvastatin reduced arterial stiffness in patients with hypertension and hypercholesterolemia, diabetes mellitus. Fassett at al. found that atorvastatin reduced arterial stiffness in CKD patients (stage 2-4) but they did not include patients on maintenance haemodialysis in their study. We want to illustrate if these beneficial effects on arterial stiffness will be present or not among haemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients on regular hemodialysis treatment for more than 3 months

Exclusion Criteria:

* Patients with diabetes mellitus.
* Patients with known severe valvular heart disease.
* Irregular heart rhythm.
* History of aortic surgery/prosthetic aorta.
* Acute liver disease.
* Patients receiving lipid lowering drugs.
* Pregnancy.
* History of myocardial infraction in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
change in Aortic pulse wave velocity (PWV) | baseline, 24 weeks
  the procedure was done at least 30 minutes after the dialysis session. Measurements were made after 10 minutes of rest in a supine position with a suitable cuff placed in the upper arm (the non-arteriovenous fistula arm in the hemodialysis group) and a connecting tube linking the cuff to a recorder device.Three consecutive measurements were taken automatically with 30 seconds of duration.
change in Augmentation index (AIx) | baseline, 24 weeks
  It is a surrogate index of arterial stiffness which measures pulse wave reflections that significantly influence the central pressure profile. It is directly related to peripheral arterial stiffness.

SECONDARY OUTCOMES:
change in Central systolic blood pressure (CSP) | 24 weeks
  Central aortic systolic blood pressure is a parameter that strongly reflects vascular changes of central elastic arteries compared to peripheral brachial blood pressure
change in Peripheral blood pressure (PBP) | baseline, 24 weeks
  change in peripheral systolic and diastolic blood pressure
change in central pulse pressure (PP) | baseline, 24 weeks
  will be clalculated from the central waveform

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; El Hassan M Ayman, MSc, Study Chair — Assistant lecturer
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stack AG, Bloembergen WE. Prevalence and clinical correlates of coronary artery disease among new dialysis patients in the United States: a cross-sectional study. J Am Soc Nephrol. 2001 Jul;12(7):1516-1523. doi: 10.1681/ASN.V1271516. PMID 11423581
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness on survival in end-stage renal disease. Circulation. 1999 May 11;99(18):2434-9. doi: 10.1161/01.cir.99.18.2434. PMID 10318666
- [Background] Chertow GM, Raggi P, Chasan-Taber S, Bommer J, Holzer H, Burke SK. Determinants of progressive vascular calcification in haemodialysis patients. Nephrol Dial Transplant. 2004 Jun;19(6):1489-96. doi: 10.1093/ndt/gfh125. Epub 2004 Apr 21. PMID 15102961
- [Background] Simionescu M. Implications of early structural-functional changes in the endothelium for vascular disease. Arterioscler Thromb Vasc Biol. 2007 Feb;27(2):266-74. doi: 10.1161/01.ATV.0000253884.13901.e4. Epub 2006 Nov 30. PMID 17138941
- [Background] Bellasi A, Ferramosca E, Ratti C. Arterial stiffness in chronic kidney disease: the usefulness of a marker of vascular damage. Int J Nephrol. 2011;2011:734832. doi: 10.4061/2011/734832. Epub 2011 May 23. PMID 21660313
- [Background] Briet M, Boutouyrie P, Laurent S, London GM. Arterial stiffness and pulse pressure in CKD and ESRD. Kidney Int. 2012 Aug;82(4):388-400. doi: 10.1038/ki.2012.131. PMID 22534962
- [Background] Adenwalla SF, Graham-Brown MPM, Leone FMT, Burton JO, McCann GP. The importance of accurate measurement of aortic stiffness in patients with chronic kidney disease and end-stage renal disease. Clin Kidney J. 2017 Aug;10(4):503-515. doi: 10.1093/ckj/sfx028. Epub 2017 May 10. PMID 28852490
- [Background] Palaniswamy C, Selvaraj DR, Selvaraj T, Sukhija R. Mechanisms underlying pleiotropic effects of statins. Am J Ther. 2010 Jan-Feb;17(1):75-8. doi: 10.1097/MJT.0b013e31819cdc86. PMID 19451808
- [Background] Sarafidis PA, Kanaki AI, Lasaridis AN. Effects of statins on blood pressure: a review of the experimental and clinical evidence. Curr Vasc Pharmacol. 2007 Apr;5(2):155-61. doi: 10.2174/157016107780368307. PMID 17430220
- [Background] Kanaki AI, Sarafidis PA, Georgianos PI, Kanavos K, Tziolas IM, Zebekakis PE, Lasaridis AN. Effects of low-dose atorvastatin on arterial stiffness and central aortic pressure augmentation in patients with hypertension and hypercholesterolemia. Am J Hypertens. 2013 May;26(5):608-16. doi: 10.1093/ajh/hps098. Epub 2013 Feb 28. PMID 23449607
- [Background] Davenport C, Ashley DT, O'Sullivan EP, McHenry CM, Agha A, Thompson CJ, O'Gorman DJ, Smith D. The Effects of Atorvastatin on Arterial Stiffness in Male Patients with Type 2 Diabetes. J Diabetes Res. 2015;2015:846807. doi: 10.1155/2015/846807. Epub 2015 Apr 30. PMID 26064990
- [Background] Fassett RG, Robertson IK, Ball MJ, Geraghty DP, Sharman JE, Coombes JS. Effects of atorvastatin on arterial stiffness in chronic kidney disease: a randomised controlled trial. J Atheroscler Thromb. 2010 Mar 31;17(3):235-41. doi: 10.5551/jat.2683. Epub 2009 Dec 24. PMID 20032570
- [Background] Wassertheurer S, Kropf J, Weber T, van der Giet M, Baulmann J, Ammer M, Hametner B, Mayer CC, Eber B, Magometschnigg D. A new oscillometric method for pulse wave analysis: comparison with a common tonometric method. J Hum Hypertens. 2010 Aug;24(8):498-504. doi: 10.1038/jhh.2010.27. Epub 2010 Mar 18. PMID 20237499
- [Background] Hametner B, Wassertheurer S, Kropf J, Mayer C, Eber B, Weber T. Oscillometric estimation of aortic pulse wave velocity: comparison with intra-aortic catheter measurements. Blood Press Monit. 2013 Jun;18(3):173-6. doi: 10.1097/MBP.0b013e3283614168. PMID 23571229
- [Derived] Elsayed MM, Ayman EM. Atorvastatin can delay arterial stiffness progression in hemodialysis patients. Int Urol Nephrol. 2022 Nov;54(11):2969-2976. doi: 10.1007/s11255-022-03231-3. Epub 2022 May 18. PMID 35585282